CLINICAL TRIAL: NCT03794622
Title: The Effect of Autologous Bone Marrow Concentration on Femoral Shaft Fracture Union
Brief Title: Autologous Bone Marrow Concentration for Femoral Shaft Fracture Union
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Pei-Yuan Lee, MD (Other)
Collaborators: Aeon Biotechnology Corporation (Industry)
Responsible Party: Sponsor-Investigator, Pei-Yuan Lee, MD, Principal Investigator, Show Chwan Memorial Hospital
Organization: Show Chwan Memorial Hospital (Other)
Other Study IDs: RD106049
Record Dates: First submitted 2019-01-02; First posted 2019-01-07 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Bone Marrow; Femoral Shaft Fracture
Keywords: Bone Marrow; Mesenchymal Stromal Cells; Femoral Shaft Fracture

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bone marrow concentration group: Consecutive patients receive intramedullary nail fixation with bone marrow concentration.
  Interventions: Other: intramedullary nail fixation with bone marrow concentration
- Historical control group: Previous age- and gender-matched patients who receive intramedullary nail fixation only.
  Interventions: Other: intramedullary nail fixation

INTERVENTIONS:
Other: intramedullary nail fixation with bone marrow concentration — intramedullary nail fixation with bone marrow concentration
  Groups: Bone marrow concentration group
Other: intramedullary nail fixation — intramedullary nail fixation only
  Groups: Historical control group

SUMMARY:
This study aims to evaluate the effect of bone marrow concentration on union of femoral shaft fracture by comparing clinical and imaging outcomes between patients receiving Intramedullary nail fixation with intraoperative bone marrow concentration and those receiving Intramedullary nail fixation only.

DETAILED DESCRIPTION:
Femoral shaft fracture is a common orthopaedic injury. Intramedullary nail is one of the standard treatments. Its primary goal is to develop an osseous bridge between adjacent motion segments to prevent motion, relieve pain, and facilitate bone union. Delayed union or nonunion is common in femoral shaft fracture. Risk factors include comminuted fracture, open fracture, smoking, diabetes and open reduction of fracture fixation. Mesenchymal stem cells are pluripotent cells that can differentiate into multiple mesenchymal tissues, including tenocytes, chondrocytes and osteoblasts, as well as being a source of multiple growth factors to establish an environment conducive to soft and hard tissue regeneration. As bone marrow concentration has high concentration of mesenchymal stem cells, some studies have shown that autologous bone marrow concentration can improve bone healing. Therefore, the goal of this study was to evaluate the effect of bone marrow concentration on union of femoral shaft fracture.

ELIGIBILITY:
Inclusion Criteria:

* With recent diagnosis of femoral shaft fracture
* Treated with intramedullary nail fixation
* With one or more risk factors of non-union: comminuted fracture, open fracture, smoking, obesity, diabetes, open reduction,
* Age between 20 and 80 years

Exclusion Criteria:

* Old femoral shaft fracture
* With concurrent major trauma, ex. intracranial hemorrhage, pneumothorax, hemothorax, internal bleeding.
* With prior history of femoral surgery
* With current or prior history of trauma or infection at femur
* With current diagnosis of coagulopathy
* With current or prior history of cancer
* With current or prior history of hematological disease
* Pregnancy
* Patients who will not cooperate with one-year followup

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive eligible patients who underwent intramedullary nail fixation combined with autologous bone marrow stem cells treatment for femoral shaft fracture
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2017-06-14 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
1-month postoperative degree of union evaluated by plain radiograph | 1-month postoperative
  Degree of union evaluated by plain radiograph

SECONDARY OUTCOMES:
2-month postoperative degree of union evaluated by plain radiograph | 2-month postoperative
  Degree of union evaluated by plain radiograph
3-month postoperative degree of union evaluated by plain radiograph | 3-month postoperative
  Degree of union evaluated by plain radiograph
6-month postoperative degree of union evaluated by plain radiograph | 6-month postoperative
  Degree of union evaluated by plain radiograph
12-month postoperative degree of union evaluated by plain radiograph | 12-month postoperative
  Degree of union evaluated by plain radiograph

CONTACTS AND LOCATIONS:
Overall Officials: Pei-Yuan Lee, MD, Study Chair — Show Chwan Memorial Hospital
Locations (1):
- Show Chwan Memorial Hospital, Changhua, Changhua, Taiwan

IPD SHARING:
Plan to Share IPD: No